CLINICAL TRIAL: NCT06725966
Title: Personalized Medicine to Treat Refractory Benign Paroxysmal Positional Vertigo, Through Computational Fluid Dynamics Analysis From Magnetic Resonance Image Reconstructions
Brief Title: Personalized Treatment of Refractory BPPV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinico Universitario de Santiago (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); European Union (Other)
Responsible Party: Principal Investigator, Andrés Soto-Varela, Professor and Chairman, Hospital Clinico Universitario de Santiago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI23/0024
Record Dates: First submitted 2024-12-02; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Benign Paroxysmal Positional Vertigo; Personalized Medicine
Keywords: BPPV; Benign paroxysmal positional vertigo; Computational fluid dynamics; MRI; Canalith repositioning maneuvers; Mechanical rotation chair
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo

STUDY DESIGN:
Intervention Model Description: Experimental, multicenter, open-label, randomized study (using balanced block randomization) with two parallel arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Epley maneuver (Active Comparator): Participants will be advised to perform Brandt-Daroff exercises at home twice daily for 8 weeks. An MRI of the inner ear and posterior cranial fossa will also be requested. If the exercises are ineffective, repositioning maneuvers using a mechanized chair will be repeated biweekly until symptom resolution.
  Interventions: Procedure: Conventional Epley maneuver
- Personalized Epley maneuver (Experimental): Participants will perform Brandt-Daroff exercises at home twice daily for 8 weeks. An MRI will be conducted, and based on the images, a personalized mathematical model will be created to modify the angles of the repositioning maneuver. If the exercises are ineffective, the personalized maneuver will be performed using a mechanized chair.
  Interventions: Procedure: Personalized Epley maneuver

INTERVENTIONS:
Procedure: Conventional Epley maneuver — Epley maneuver using a mechanized chair
  Arms: Conventional Epley maneuver
Procedure: Personalized Epley maneuver — Personalized Epley maneuver, using a mechanized chair
  Arms: Personalized Epley maneuver

SUMMARY:
Background: Benign paroxysmal positional vertigo (BPPV) is the most common cause of vertigo, often effectively treated with standard canalith repositioning maneuvers (CRMs). However, approximately 12.5% of cases remain refractory, leading to persistent symptoms and increased healthcare burden. Variations in the anatomical orientation of the semicircular canals (SCCs) may explain the resistance to conventional maneuvers. This study explores a personalized medicine approach, utilizing computational fluid dynamics (CFD) based on MRI reconstructions to tailor CRMs with the help of mechanical rotation chair according to individual inner ear anatomy.

Methods: The investigators conducted a randomized, multicenter, open-label study targeting patients with refractory posterior canal BPPV. Participants were allocated to either a control group (receiving repeated standard CRMs and Brandt-Daroff exercises) or an intervention group (receiving personalized CRMs based on CFD simulations derived from MRI scans). The intervention group's maneuvers were executed using a mechanical rotational chair designed for precise angulation. Primary outcomes included resolution of nystagmus and vertigo symptoms, while secondary outcomes measured the reduction in healthcare visits and improved quality of life (Dizziness Handicap Inventory score).

DETAILED DESCRIPTION:
1. STUDY DESIGN This is an experimental, multicenter, open-label, randomized study (using balanced block randomization) with two parallel arms. The study targets patients with a definitive diagnosis of refractory posterior semicircular canal BPPV (BPPVp).
2. STUDY PARTICIPANTS Study Period: From January 1, 2024, to December 31, 2026. Study Population: Patients diagnosed with BPPV. Target Population: Individuals >18 years of age, of both sexes, diagnosed with unilateral refractory BPPVp, from three Health Areas. Participants will be selected from patients attending the Otoneurology Unit of the Otolaryngology Departments of these three University Hospital Complexes.

   To confirm the diagnosis and rule out other potential causes, all participants will undergo a complete otoneurological evaluation, including:
   * Otoscopy.
   * Basic neurological examination.
   * Observation of spontaneous nystagmus (with and without gaze fixation).
   * Clinical head impulse test (vHIT), including video-assisted evaluation.
   * Positional tests (DHT, McClure test, and head hyperextension), with videonystagmographic recording.
   * Pure-tone audiometry. In cases of refractory BPPV (lack of resolution after three therapeutic maneuvers), a magnetic resonance imaging (MRI) scan of the inner ears and posterior cranial fossa will be requested to rule out central neurological causes.
3. RANDOMIZATION

   Pre-selection Visit (Visit -1): Participants will undergo a comprehensive vestibular assessment to identify candidates with refractory BPPVp. The following tests will be included:
   * Video-assisted head impulse test (vHIT) to assess for other vestibular pathologies.
   * Dix-Hallpike test (DHT) to confirm the diagnosis of BPPVp.
   * McClure test to exclude horizontal canal BPPV.
   * Head hyperextension test to exclude superior canal BPPV.
   * Dizziness Handicap Inventory (DHI) questionnaire adapted to Spanish, assessing perceived disability due to vertigo.

   For posterior canal BPPV, it will be verified in the medical record that three repositioning maneuvers (Epley and/or Semont) were performed without symptom resolution.

   Eligible participants will be given a detailed explanation of the study objectives and procedures, and will receive the approved Patient Information Sheet (PIS) to provide informed consent.
4. RANDOMIZATION PROCESS

   Visit 0 (Randomization Visit): After obtaining consent, participants will be randomized to one of the following study arms:

   • Control Group: Participants will be advised to perform Brandt-Daroff exercises at home twice daily for 8 weeks. An MRI of the inner ear and posterior cranial fossa will also be requested. If the exercises are ineffective, repositioning maneuvers using a mechanized chair will be repeated biweekly until symptom resolution.

   • Study Group: Participants will perform Brandt-Daroff exercises at home twice daily for 8 weeks. An MRI will be conducted, and based on the images, a personalized mathematical model will be created to modify the angles of the repositioning maneuver. If the exercises are ineffective, the personalized maneuver will be performed using a mechanized chair.

   A balanced block randomization sequence with block size n=10 will be generated by a member of the research team.
5. DATA COLLECTION

   Even if intermediate visits are necessary, the following study visits will be conducted according to the protocol (with data recording):
   * Visit 1 (Eight Weeks After Inclusion):

     - The Dix-Hallpike Test (DHT) will be performed with videonystagmographic recording. If positive:

     - In the control group, the conventional Epley maneuver will be repeated using a mechanized chair.
     * In the study group, a personalized Epley maneuver will be performed using a mechanized chair.
   * Visit 2 (Ten Weeks After Inclusion):

     * The DHT will be repeated with videonystagmographic recording. If positive:
     * In the control group, the conventional Epley maneuver will be repeated using a mechanized chair.
     * In the study group, the personalized Epley maneuver will be repeated using a mechanized chair.

   These maneuvers (conventional for the control group and personalized for the study group) will be repeated every two weeks until resolution of symptoms (or up to a maximum of 8 repetitions).

   • Visit 3 (Six Months After Inclusion):

   - The following variables will be recorded:

   - Dix-Hallpike Test (DHT) results (negative or positive).
   * Dizziness Handicap Inventory (DHI) score.
   * Number of consultations required for resolution.

5. MATHEMATICAL STUDY A 3D model of the affected membranous labyrinth will be reconstructed based on MRI imaging. An analysis of the planes on which the semicircular canals rest will be performed, and the geometric model will be adapted for subsequent numerical simulation. The computational study, carried out using Computational Fluid Dynamics (CFD) techniques, will involve combining the dynamics of the endolymph within the labyrinth and the particle dynamics of the free otoliths.

Mathematically, the Navier-Stokes equations will be coupled with a discrete particle model sensitive to gravity and the fluid forces. This will allow for the determination of the velocity distribution of the endolymph, the pressures exerted on the labyrinth walls, as well as the timing and positions of the otoliths during the personalized Epley maneuver.

6. DATA ANALYSIS Demographic data and patient characteristics will be described globally and by relevant covariables.

Continuous outcomes will be summarized using mean, median, standard deviation (SD), and interquartile range (P25, P75). For categorical outcomes, the number and percentage of patients in each category will be reported. Statistical analyses will be based on the full analysis set (FAS), which includes all randomized participants who provided informed consent and met all inclusion criteria without any exclusion criteria.

7. STUDY LIMITATIONS, DATA BIASES, AND MITIGATION STRATEGIES Despite being an open-label study, the potential bias introduced is minimal, as both the maneuvers and outcome evaluation are performed by the same person. The primary outcome (resolution of nystagmus) is assessed objectively through videonystagmography, which does not require interpretation by the evaluator.

There is a risk of patient dropout during the eight-week period of Brandt-Daroff exercises prior to the personalized maneuver. To mitigate this risk, patient adherence will be closely monitored and encouraged.

Since patients will be recruited from three different hospitals, there may be diagnostic biases depending on the evaluator. However, all intervention maneuvers (both personalized and conventional) will be conducted at a single center, where a diagnostic reevaluation will be performed prior to intervention to confirm that the BPPV remains unresolved and exclusively affects the posterior canal.

8. SAMPLE SIZE AND CALCULATION METHODOLOGY To estimate the sample size, the investigators assume that approximately 25% of patients with refractory BPPVp may be cured through repeated maneuvers or Brandt-Daroff exercises (control group). A significant difference of 50% in the study group (i.e., a 75% efficacy rate for symptom resolution) is considered clinically meaningful. With a 95% confidence level (1-α) and 95% statistical power for a two-tailed hypothesis test, a sample size of 23 participants per arm is required. Thus, the estimated total sample size is 46 individuals, increased to 54 (27 per group) to account for a 15% anticipated dropout rate.

ELIGIBILITY:
Inclusion Criteria:

* A. Diagnosed with BPPVp according to the Barany Society criteria:

  1. Recurrent episodes of vertigo or positional instability, triggered by lying down or turning the head in the supine position.
  2. Episodes lasting less than 1 minute.
  3. Positional nystagmus observed after a latency period during the Dix-Hallpike test (DHT), with an upward vertical component and a torsional component (clockwise on the left side and counterclockwise on the right).
  4. Symptoms not explained by any other cause.

     AND
* B. Refractory to otolith repositioning maneuvers (Epley and/or Semont maneuvers), with persistence of symptoms after three attempts.

Exclusion Criteria:

* Cognitive impairment that prevents understanding of their condition and the required procedures.
* Pathological conditions that hinder the execution of the maneuvers.
* BPPV involving canals other than the posterior canal or bilateral posterior canal involvement.
* Low educational level, which may impede understanding of the procedures and informed consent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of curation | 6 months
  Percentage of participants in whom, after the maneuvers, no nystagmus is observed in the Dix and Hallpike test

SECONDARY OUTCOMES:
Rate of resolution of symptomatology | 6 months
  Percentage of participants who, after the maneuvers, do not report vertigo in the Dix and Hallpike test
DHI score | 6 months
  DHI (Dizzines Handicap Inventory) score after the maneuvers, compared to the score at the time of inclusion
Number of sessions | 6 months
  Number of maneuvers need to curation

CONTACTS AND LOCATIONS:
Overall Officials: Andrés Soto-Varela, Prof, PhD, Principal Investigator — Complexo Hospitalario Universitario de Santiago
Locations (1):
- Hospital Clínico Universitario, Santiago de Compostela, A Coruña, Spain

REFERENCES:
- [Derived] Rossi-Izquierdo M, Santos-Perez S, Aran-Tapia I, Blanco-Ulla M, Aran-Gonzalez I, Vaamonde-Sanchez-Andrade I, Franco-Gutierrez V, Perez-Munuzuri V, Munuzuri AP, Soto-Varela A. Personalized medicine to treat refractory benign paroxysmal positional vertigo, through computational fluid dynamics analysis from magnetic resonance image reconstructions. Front Neurol. 2025 Mar 11;16:1561356. doi: 10.3389/fneur.2025.1561356. eCollection 2025. PMID 40134694